CLINICAL TRIAL: NCT02308241
Title: A Pilot Study of Ribavirin for Patients With Recurrent/Metastatic (R/M) Human Papillomavirus (HPV)-Related Malignancies
Brief Title: Ribavirin for Patients With Recurrent/Metastatic (R/M) Human Papillomavirus (HPV)-Related Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-211
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-03

CONDITIONS: Human Papillomavirus (HPV)-Related Malignancies; Recurrent/Metastatic (R/M) Human Papillomavirus (HPV)-Related Malignancies
Keywords: Ribavirin; Human Papillomavirus (HPV); Recurrent/Metastatic (R/M); 14-211
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Ribavirin

ARMS (1):
- Ribavirin (Experimental): Study subjects will self-administer ribavirin 1400 mg PO BID (total dose, 2800 mg/day). All patients will complete pill diaries to document administration of study drug. Cycle length is 28 days with continuous dosing. Clinic visits for safety assessments and routine laboratory studies will occur weekly in Cycle 1, in weeks 1 and 3 of Cycle 2, and on Week 1 of subsequent cycles. Cross sectional imaging (CT or MRI) is obtained at baseline and q2 cycles and at End-of Treatment (EOT). Response assessments will follow RECIST 1.1 criteria.
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — self-administer ribavirin 1400 mg PO BID (total dose, 2800 mg/day)

SUMMARY:
The purpose of this study is to find out the effects, both good and bad, that a drug called ribavirin has on the patient and the cancer.

Ribavirin has also been studied in clinical trials for patients with various types of cancer. These studies demonstrated that ribavirin can be safely given at higher doses than the dosing that is used as part of the treatment of hepatitis C.

Ribavirin is known to target a protein called "4E" that turns on a central part which causes the cell to grow, called the ribosome. HPV-related cancers often have abnormally high levels of 4E. The purpose of this study is to evaluate if ribavirin may be a useful treatment for patients with advanced cancers that are related to HPV by blocking the activity of 4E.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent and/or metastatic HPV-related carcinoma of the cervix, anus, vagina, vulva, penis, or oropharynx. The cancer diagnosis must be confirmed by slide review in the MSKCC Department of Pathology. HPV positive status must be demonstrated by HPV in situ-hybridization (ISH) and/or by p16 immunohistochemistry (IHC).

Note: For cervix squamous cancer, HPV ISH test or p16 IHC test is not required, because all cervix squamous cancers are presumed to be HPV-associated.

* Adults (≥ 18 years of age)
* ECOG performance status of 1 or better
* Measurable disease according to RECIST 1.1 criteria
* Availability of archived tumor tissue for correlative studies (5 unstained slides)
* Adequate organ function, as follows:
* Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 X 109/L, platelets ≥ 160 X 109/L, hemoglobin ≥ 10 g/dL
* Hepatic: total bilirubin within ULN (upper limit of normal); alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.0 X ULN
* Renal: Serum creatinine ≤ 1.3 mg/dL. Patients with serum creatinine > 1.3 mg/dL may be eligible if creatinine clearance (CrCl) ≥ 55 mL/min based on the standard Cockroft and Gault formula.
* Ability to swallow oral medication.
* Patients of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Patients must agree to use a reliable method of birth control during and for 6 months following the last dose of study drug.
* At least one prior systemic therapy regimen for R/M HPV-related carcinoma

Exclusion Criteria:

* History of hemolytic anemia or thalassemia
* Current treatment or known prior treatment with ribavirin
* Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment.
* Current therapeutic anticoagulation with Coumadin (warfarin)
* Known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- [Derived] Burman B, Drutman SB, Fury MG, Wong RJ, Katabi N, Ho AL, Pfister DG. Pharmacodynamic and therapeutic pilot studies of single-agent ribavirin in patients with human papillomavirus-related malignancies. Oral Oncol. 2022 May;128:105806. doi: 10.1016/j.oraloncology.2022.105806. Epub 2022 Mar 23. PMID 35339025
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ribavirin
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ribavirin
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 59 [47 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Responses, Determined by RECIST 1.1 Criteria
Description: will be tabulated by adding partial responses and complete responses (CR + PR). The regimen would be considered worthy of further study if radiographic responses are observed in at least 2 of 12 subjects.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin
Number analyzed (Participants) | 12
Participants
  Stable Disease | 5
  Progression of Disease | 4
  Unevaluable | 3

2. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: will be tabulated using NCI CTCAE version 4,
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ribavirin
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin (N=12)
Anemia (Blood and lymphatic system disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Blood bilirubin increased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Aspartate aminotransferase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
Fever (General disorders) | 3
White blood cell decreased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
INR increased (Investigations) | 2
Investigation - Other, specify (Investigations) | 2
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Paronychia (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT02308241/Prot_SAP_000.pdf